CLINICAL TRIAL: NCT06025097
Title: Therapeutic Effect of Intra-Tympanic Methyl Prednisone-platelet Rich Plasma Combination in Sensorineural Hearing Loss and Tinnitus of Cochlear Origin.
Brief Title: Intra-Tympanic Steroid With PRP Combination in Sensorineural Hearing Loss and Tinnitus.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CMH RWP Combined Military Hospital RWP: Rawalpindi (Other Government)
Responsible Party: Principal Investigator, Muhammad Noman Karim, Principal Investigator, Otolaryngology Dept, CMH Rawalpindi, CMH RWP Combined Military Hospital RWP: Rawalpindi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2023-08-10; First posted 2023-09-06 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Sensorineural Hearing Loss; Tinnitus
Keywords: Steroids; Platelet rich plasma; intratympanic steroids
MeSH Terms: conditions — Hearing Loss, Sensorineural; Tinnitus | interventions — TEC solution; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Intervention Model Description: Single group study, to show the therapeutic effects of Combination solution on diseases in fixed time.
Masking Description: Care giver and patient both are known to the treatment being offered under investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Treated Arm (Experimental): Single arm study, Patients with SNHL and Tinnitus all were given same Composite solution consisting of (Methyl prednisone and Platelet rich plasma) via intr-atympanic route..
  Interventions: Drug: Combination Solution

INTERVENTIONS:
Drug: Combination Solution — Methyl Prednisone (Trade name: SOLU-MEDROL) + Platelet rich Plasma (Autologous Biological product) via intra-tympanic rout about 1-1.5 ml.
  Other Names: PRP + Solumedrol

SUMMARY:
Steroids are used widely for the treatment of Sensorineural hearing loss worldwide. The difficulty lies with efficient delivery of the drug into the cochlea, which is already a sealed chamber with limited blood supply that too with an end Artery. We intend to extrapolate its effects by combining it with Platelet rich plasma. intra-tympanic delivery is achieved with injection via tympanic membrane and its absorption via round window is hastened by posture maintenance for about half an hour. PRP is an autologous biologic fluid which has excellent safety profile and is already in use by various specialties.

DETAILED DESCRIPTION:
Definitions:

Sensorineural Hearing Loss: Hearing loss occurring due to pathologies of cochlea.

Platelet-rich plasma : Platelet-rich plasma is an autologous biological product separated from blood after removal of Red blood cells. It is the plasma portion of blood which is simply rich of platelets.

Preparations:

Intratympanic methyl prednisone + Autologous PRP: 2ml Solution (1ml of methyl prednisone 40mg/ml + 1ml of PRP)

Materials and Methods:

Inclusion Criteria:

mentioned in pertinent section

Exclusion Criteria:

mentioned in pertinent section

Methodology:

This will be an Interventional study, prior permission from Hospitals Ethical Review Board will be taken. Informed consent will be obtained from the patients with regards to participation the study. All the patients in which the presentation to Ear Nose Throat (ENT) clinic is SNHL or Subjective tinnitus and also satisfying the inclusion criteria will be selected. SNHL will be graded according to the audiogram and values will be recorded to the nearest +5db with round off. The Tinnitus will be graded on visual analogue scale graded from 1 to 10 (1= No tinnitus while 10 being the worst). After recording the pre-treatment data these patients will be scheduled for intervention. Patients will receive the solution consisting of 1ml methyl prednisone (40mg/ml) and 1ml of PRP via intra-tympanic route. The solution will be injected into the tympanic cavity via the tympanic membrane injection (intra-tympanic route). Patients will receive repeated doses of same intra-tympanic injections on every third day for a total of 3 consecutive doses (in 9 days). Hearing assessment via Audiometry will be done post-treatment after 2 weeks of finishing the treatment (23rd day after starting the therapy).

Procedure: On receiving a patient at ENT department with a diagnosis of SNHL/ tinnitus, patient will be scheduled for intra-tympanic injection session. All of the intra-tympanic injections will be performed by the same ENT Doctor. Patient will be positioned in sitting posture, head tilted sideways and rotated slightly to instill the pyodine solution into the ear for 5 minutes. Then after cleaning with a sterile suction tip, xylocaine 10% solution will be sprayed into the ear canal and a wick soaked in xylocaine left there for 5 more minutes. The wick will then be removed and ear will be examined to exclude any physical disease or deformity in the external ear. Head will be brought to the examining position and a sterile 3cc syringe will be loaded with 1 ml of 40mg/ml methyl prednisone and 1 ml of PRP. 3cc syringe needle is replaced with 25 Guage Lumber Puncture needle. Under guidance of a Microscope or 0-degree rigid Endoscope, one point Pin-hole will be made by just piercing the Tympanic membrane antero-inferiorly and the prepared solution will be instilled. While instilling the solution a meniscus would be seen rising from inferior to superior aspect of the tympanic membrane. The patient will be made to lie in supine position and then will be made to stay in same position for about 15-30 mins (so as to hasten the absorption through round window and to prevent escape of solution via Eustachian tube). This supine position would also facilitate establishment of a reservoir in the mastoid antrum to slowly discharge over time and further the absorption through round window. A cotton wick will be left in the ear canal to be removed after an hour. The procedure will be repeated at every 3rd day till a total of three procedures. Patient will be further called for follow up Audiometry, at 2 weeks after finishing the treatment. Any improvement from the pre-treatment audiometry will be noted. Improvement will be labelled as Mild; of 10 decibels, partial; 11-25 decibels and Good; above 25 decibels. The improvements in tinnitus will be ascertained subjectively with a visual analogue scale graded from 1 to 10. Data will be recorded and analyzed and results will be published in due course of time.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10-70 yrs
* Capacity to have a Pure tone Audiometry test
* Disease

  1. SNHL;

     * Unilateral or bilateral sensorineural hearing loss
     * Without any identifiable cause
  2. Tinnitus;

     * Subjective sensation of noise without any obvious source of sound
     * Without any identifiable cause
* Hearing levels of 55dB or above

Exclusion Criteria:

* Age: less than 10 or more than 70 yrs
* Conductive hearing loss/ Mixed Hearing loss
* Tumor, Neurologic cause of hearing loss/ tinnitus
* Past ear Surgery
* Any External, middle or inner Ear Disease other than SSNHL
* Traumatic Hearing Loss or Hearing Loss due to an obvious cause.
* Patients' refusal to follow-up
* Any contraindication to Steroids administration.
* Any Blood Disorder
* Non-consenting patients
* Comorbid:

  * Diabetes
  * Hypertension
  * Cardio vascular diseases
  * Obesity
  * Etc.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-21 (Actual)

PRIMARY OUTCOMES:
Improvement in Hearing | 2 weeks post treatment completion.
  Improvement in hearing as per Audiogram, measured in decibels.
Improvement in Tinnitus | 2 weeks post treatment completion.
  Improvement in Tinnitus as per Visual analogue scale from 1 to 10 with 1 being the lowest improvement and 10 being the best.

CONTACTS AND LOCATIONS:
Overall Officials: Farhan Akbar, FCPS, Study Director — CMH Rawalpindi
Locations (1):
- Combined Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
If there is a need to analyze the data for a particular clinical question, than only the data would be shared with other researchers.